CLINICAL TRIAL: NCT03755167
Title: An Open-Label, Multi-Center, Follow up Study to Protocol 101/2 - Continued Treatment by Intravenously Administered IPL344 to Amyotrophic Lateral Sclerosis (ALS) Patients
Brief Title: A Follow up Study to Protocol 101/2 - Continued Treatment by IPL344 IV
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was suspended due to IPL344 shortage and may resume once drug supply is available. Survival follow-up is still ongoing following participants' consent
Sponsor: Immunity Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101/3
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPL344 (Experimental): IV IPL344 administered once a day
  Interventions: Drug: IPL344

INTERVENTIONS:
Drug: IPL344 — IPL344 will be administered by intravenously (IV) infusion once a day (every 24±6 hours), using a Peripherally Inserted Central Catheter (PICC) line or a permanent port. IPL344 will be administered using an electronic pump at a flow rate that will be determined in protocol 101/2. The dose will be fixed as MTD as established in protocol 101/2 (up to 3.2 mg/kg).

SUMMARY:
This is a prospective, open-label, follow up study to protocol 101/2 - continued treatment by IPL344 IV administered once a day in up to 15 participants with ALS.

The study is designed to determine the safety, tolerability and initial efficacy of IPL344, administered once a day, by IV infusion for up to 36 months

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ages ≥ 18 to 75 years.
2. Participants that have completed study protocol #101/2
3. A written informed consent signed prior to any study procedure being performed
4. Medically capable to undergo study procedures at the time of study entry

Exclusion Criteria:

1. Participants that did not participate or did not complete 28 treatment days of study protocol #101/2.
2. Concurrent therapy, that in the PI's opinion, would interfere with the evaluation of the safety or efficacy of the study medication
3. Presence of any other condition or circumstance that, in the judgment of the Investigator, might contraindicate or increase the risk to the participant.
4. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative serum pregnancy test from protocol 101/2)
5. Women of child-bearing potential or males whose partners are women of child-bearing potential, unwilling or unable to use an effective method of contraception throughout the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-12-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) Reporting | upto 36 month
  All AEs will be recorded, whether considered minor or serious, drug-related or not

SECONDARY OUTCOMES:
Changes from baseline in ALS disease progression | upto 36 months
  Evaluated by the Amyotrophic Lateral Sclerosis Functional Rating Scale(ALSFRS-R). The ALSFRS-R is a quickly administered (5 min) ordinal rating scale used to determine a subject's assessment of their capability and independence in 12 functional activities. There are 12 questions, graded by the subject 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects speech and swallowing, fine motor skills, large motor skills, and breathing

OTHER OUTCOMES:
Changes from baseline in Pulmonary Function | upto 36 months
  Measured by Vital Capacity (VC)
Changes from baseline in Muscle strength | upto 36 months
  Assessed by using a quantitative strength testing tool, Hand Held Dynamometry (HHD)
Changes from baseline in Muscle strength | upto 36 months
  Assessed by using a quantitative strength testing tool - hand grip
Changes from baseline in Anti-Depression effect | upto 36 months
  Evaluated by ALS Depression Inventory (ADI-12). Scales: For each question, the following is selected: "I fully agree", "I agree", "I don't agree", "I do not agree at all"
Changes from baseline in Anti-Depression effect | upto 36 months
  Evaluated by the Hospital Anxiety and Depression Scale (HADS). The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Hadassah Medical Center/Neuromuscular / EMG service and ALS / Motor Neuron Disease Clinic, Jerusalem
  - Hadassah Medical Center -Motor Neuron Disease Clinic, Jerusalem

IPD SHARING:
Plan to Share IPD: Undecided